CLINICAL TRIAL: NCT01818765
Title: Left Ventricular Endocardial Pacing Through the Ventricular Septum
Brief Title: A Pilot Study of Interventricular Septal Puncture for Cardiac Resynchronization Therapy to Treat Heart Failure
Acronym: LV-CONSEPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Heart Research UK (Unknown)
Responsible Party: Principal Investigator, Dr James Gamble, Co-Investigator, Oxford University Hospitals NHS Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OUH-2013-208; 13/SC/0186 (Other: United Kingdom National Research Ethics Service)
Record Dates: First submitted 2013-03-19; First posted 2013-03-26 (Estimated); Results first posted 2019-10-23 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Heart Failure
Keywords: Cardiac resynchronisation therapy; Endocardial; Pacing
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Procedure (Experimental): Pre-procedure speckle-tracking echocardiography assessment of latest activation
  Trans-ventricular-septal placement of LV pacing lead
  Acute response assessment
  Interventions: Procedure: Trans-ventricular-septal placement of LV pacing lead; Other: Pre-procedure speckle-tracking echocardiography; Other: Acute response assessment

INTERVENTIONS:
Procedure: Trans-ventricular-septal placement of LV pacing lead
Other: Pre-procedure speckle-tracking echocardiography — Assessment of site of latest mechanical activation
Other: Acute response assessment — Cardiac output monitoring

SUMMARY:
Cardiac resynchronization therapy (CRT) is known to result in significant improvement in the symptoms of selected patients with heart failure, and to reduce hospital admission and death rates in these patients. CRT can improve cardiac function by improving the coordination of the heart beat using a special pacemaker. This requires a wire in the coronary sinus, one of the veins running around the outside of the heart, to stimulate the outside of the left ventricle (main pumping chamber).

There are two particular issues with this standard technique. In some patients it is not possible to get the wire into the coronary sinus due to difficult vein shapes, and in others the wire can be put there, but it does not end up in a suitable position to act on the heart enough to improve heart function. This is thought to be a major part of the reasons why one in four patients does not improve with CRT ("non-responders").

The investigators have developed a novel method of pacing the left ventricle of the heart by putting the wire through a tiny hole made in the muscle between the left and right ventricles and pacing the inside surface of the left ventricular chamber. This will allow patients in whom the coronary sinus cannot be used to have CRT. The investigators will also offer it to patients who have not improved with CRT, as there is evidence that they may respond to this procedure due to physiological benefits from pacing the inside rather than the outside and also the ability to steer the lead anywhere on the inner surface.

The investigators have performed this new procedure in a small number of patients already. This study will allow closer follow-up of more patients, and also investigation of ways to optimize results of the procedure for these patients.

DETAILED DESCRIPTION:
CRT as a treatment for heart failure in selected patients has been shown to decrease both hospitalizations and mortality as well as improving symptoms and quality of life, and is hence supported by guidelines including NICE (United Kingdom National Institute for clinical excellence) . It is achieved by placing a lead to pace the epicardial left ventricle (LV) via the coronary sinus and a coronary vein. Unfortunately, in 5-8% of patients the LV lead cannot be delivered and in 15-20% the lead is placed in a suboptimal position due to the presence of left ventricular scarring, phrenic nerve stimulation or adverse coronary vein anatomy. After lead delivery, 20-45% of patients undergoing CRT fail to respond to their implant. Suboptimal lead position is thought to be one of the most significant causes of non-response.

In the case of failed lead placement there are no well-established alternatives. The most common solution is open-chest surgery using a thoracotomy to place a lead on the epicardial surface of the heart, a procedure with considerable morbidity and a risk of death. Given the co-morbidity profile of patients suitable for CRT, and their severe heart failure, many patients are not fit enough for surgical lead placement. An alternative approach is a percutaneous procedure passing the lead through a puncture in the inter-atrial septum and across the mitral valve, in order to pace the endocardial surface of the left ventricle. This is achieved in a complex and technically-challenging procedure using both femoral and subclavian venous access. This approach exposes a long segment of lead to the systemic circulation, particularly in the low-pressure, low-flow left atrium, raising the thromboembolic risk. It can also worsen mitral regurgitation and exposes the mitral valve to a risk of damage and incompetence should lead extraction be required.

Recent studies have suggested that LV endocardial pacing offers a number of physiological advantages over the conventional epicardial approach. The lead can be positioned at any site on the endocardial surface, away from scar tissue and the phrenic nerve and at the site of maximal haemodynamic improvement, rather than being limited by venous anatomy, thus improving response to CRT. There is also evidence that endocardial pacing may of itself improve haemodynamics to a greater extent than epicardial pacing, in both animal models and in acute haemodynamic studies in humans, and provide a more physiological mechanism of activation, which may be less arrhythmogenic. Consistent with this, response to CRT with endocardial pacing in patients who had not responded to epicardial CRT has been reported, and response rates in previous reports of LV endocardial pacing have been high at approximately 90%.

Targeting of CRT lead placement is an important factor and multiple techniques have been investigated. Targeting of lead placement guided by the site of latest mechanical activation assessed with speckle-tracking echocardiography has been shown to increase response and improve long-term clinical outcomes. Anatomy limits epicardial lead positioning and the best outcomes were obtained in the 60% of patients with a lead able to be placed in the optimal site4. Cardiac output monitoring used to guide lead placement maximizes cardiac output achieved and increases the frequency of long term improvement in cardiac function. Electrical mapping can identify the site of latest electrical activation, although there is not yet evidence as to whether guiding lead position with this improves clinical outcomes. No comparisons between these techniques have been performed.

There is little published so far on how to optimize lead positioning for endocardial LV leads. Groups have so far used invasive cardiac output monitoring to assess the best position for endocardial leads, and have shown that this optimizes cardiac output at the time of implant. Despite the best available evidence for guiding conventional LV lead positioning supporting speckle-tracking echocardiography, this has not yet been used for guiding endocardial lead positioning.

The investigators propose to investigate a novel LV endocardial pacing technique using a puncture through the inter-ventricular septum. This technique has been developed and used in Oxford for a small number of patients, with an initial case series soon to be submitted for publication. Potential advantages include that the inter-ventricular septum is punctured from the same subclavian vein access site through which the other leads are inserted, and that the dilated left ventricular cavity provides a large target, reducing complications. Furthermore, lead placement and extraction would not risk damage to the mitral valve.

All patients who have a left ventricular endocardial pacing lead implanted should be anticoagulated to minimize the risk of stroke from systemic thromboembolism. It has previously been shown that most lead thrombi arise on (right) atrial leads. The investigators' study technique would allow LV endocardial pacing with no lead in the left atrium, likely reducing thromboembolic stroke risk. It is likely that a significant proportion of patients eligible for this study will already be on warfarin due to prior atrial fibrillation or other indications.

Over the last 12 months the investigators have used this novel technique on 6 patients, all of whom had an LV lead safely delivered without complication. Having refined the technique, this Phase 2 study aims to assess the feasibility and safety of the procedure in a larger cohort of patients as well as documenting echocardiographic, biochemical, and functional response.

The population under study would be two groups: firstly, patients with conventional indications for CRT who are not able to have lead implantation via the normal coronary sinus route due to adverse anatomy revealed during a failed prior attempt; and secondly, patients with a successful conventional CRT lead placement who have not responded to the therapy (non-responders). Patients with a failed lead implantation would previously either have been considered for surgical epicardial lead implantation or left with no CRT device. Non-responders are also assessed for surgical lead implantation if they are felt to be likely to respond.

No single technique is known to define optimal lead positioning, and accordingly the investigators intend to use multiple techniques to try and optimize lead positioning, both to try and find the optimal site for each patient, and to allow for comparisons between them. This would include speckle-tracking echocardiography before the procedure, as well as electrical mapping of the LV activation pattern and cardiac output monitoring during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Participants with standard indications for CRT AND
* Unable to position a LV lead via the standard coronary sinus route OR
* Non-responder to conventional CRT

Exclusion Criteria:

* Patients in whom, in the opinion of the investigators, an alternative route for LV lead placement would be safer or more effective for the patient
* Contraindications to oral anticoagulation or inability to safely take oral anticoagulation.
* Female participants who are pregnant, lactating or planning pregnancy during the course of the study.
* Participant who is terminally ill
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Betts, MBChB, Principal Investigator — Oxford University Hospitals
Locations (1):
- Oxford University Hospitals NHS Trust, Oxford, United Kingdom

REFERENCES:
- [Background] Gamble JH, Bashir Y, Rajappan K, Betts TR. Left ventricular endocardial pacing via the interventricular septum for cardiac resynchronization therapy: first report. Heart Rhythm. 2013 Dec;10(12):1812-4. doi: 10.1016/j.hrthm.2013.07.033. Epub 2013 Jul 23. No abstract available. PMID 23891954
- [Background] Bordachar P, Derval N, Ploux S, Garrigue S, Ritter P, Haissaguerre M, Jais P. Left ventricular endocardial stimulation for severe heart failure. J Am Coll Cardiol. 2010 Aug 31;56(10):747-53. doi: 10.1016/j.jacc.2010.04.038. PMID 20797486
- [Background] Khan FZ, Virdee MS, Palmer CR, Pugh PJ, O'Halloran D, Elsik M, Read PA, Begley D, Fynn SP, Dutka DP. Targeted left ventricular lead placement to guide cardiac resynchronization therapy: the TARGET study: a randomized, controlled trial. J Am Coll Cardiol. 2012 Apr 24;59(17):1509-18. doi: 10.1016/j.jacc.2011.12.030. Epub 2012 Mar 7. PMID 22405632
- [Background] Khan FZ, Virdee MS, Gopalan D, Rudd J, Watson T, Fynn SP, Dutka DP. Characterization of the suitability of coronary venous anatomy for targeting left ventricular lead placement in patients undergoing cardiac resynchronization therapy. Europace. 2009 Nov;11(11):1491-5. doi: 10.1093/europace/eup292. PMID 19880411
- [Background] Spragg DD, Dong J, Fetics BJ, Helm R, Marine JE, Cheng A, Henrikson CA, Kass DA, Berger RD. Optimal left ventricular endocardial pacing sites for cardiac resynchronization therapy in patients with ischemic cardiomyopathy. J Am Coll Cardiol. 2010 Aug 31;56(10):774-81. doi: 10.1016/j.jacc.2010.06.014. PMID 20797490
- [Background] Pratola C, Notarstefano P, Toselli T, Artale P, Squasi P, Baldo E, Ferrari R. Noncontact mapping of left ventricle during CRT implant. Pacing Clin Electrophysiol. 2010 Jan;33(1):74-84. doi: 10.1111/j.1540-8159.2009.02578.x. Epub 2009 Oct 10. PMID 19821940
- [Background] Ginks MR, Shetty AK, Lambiase PD, Duckett SG, Bostock J, Peacock JL, Rhode KS, Bucknall C, Gill J, Taggart P, Leclercq C, Carr-White GS, Razavi R, Rinaldi CA. Benefits of endocardial and multisite pacing are dependent on the type of left ventricular electric activation pattern and presence of ischemic heart disease: insights from electroanatomic mapping. Circ Arrhythm Electrophysiol. 2012 Oct;5(5):889-97. doi: 10.1161/CIRCEP.111.967505. Epub 2012 Jul 25. PMID 22832673
- [Background] Betts TR, Gamble JH, Khiani R, Bashir Y, Rajappan K. Development of a technique for left ventricular endocardial pacing via puncture of the interventricular septum. Circ Arrhythm Electrophysiol. 2014 Feb;7(1):17-22. doi: 10.1161/CIRCEP.113.001110. Epub 2014 Jan 14. PMID 24425419
- See also: UK NIHR Oxford Biomedical Research Centre — http://oxfordbrc.nihr.ac.uk/

RESULTS

PARTICIPANT FLOW:
Groups:
- Procedure: 20 patients were recruited, 15 with failed transvenous LV (left ventricular) lead placement and 5 non-responders to CRT (cardiac resynchronisation therapy) .
Period: Overall Study
Arm/Group | Procedure
Started | 20
Completed (Assessed at 6 months) | 18
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Groups:
- Procedure: 20 patients were recruited, 15 with failed transvenous LV lead placement and 5 non-responders to CRT.
Arm/Group | Procedure
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 16
Region of Enrollment [Number; unit: participants]
  United Kingdom | 20
Electrocardiogram QRS segment duration [Mean (Standard Deviation); unit: ms] | 157 (14)
ischaemic aetiology [Count of Participants; unit: Participants] | 9
Ejection fraction [Mean (Standard Deviation); unit: % (of blood ejected from left ventricle)] | 28 (7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Free of Adverse Effects at 6 Months Post Procedure
Description: Acute: coronary arterial damage; tamponade or effusion; acute lead displacement; peri-procedural systemic thromboembolism; arrhythmia; bleeding
  Chronic: systemic thromboembolism; lead displacement, dysfunction or fracture; system infection; bleeding; arrhythmia; death
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Procedure
Number analyzed (Participants) | 20
Participants | 15

2. Secondary Outcome: Procedural Success - Number of Participants With Successful Delivery of Left Ventricular Lead Via Ventricular Transseptal Approach
Description: Ability to successfully deliver LV endocardial pacing via the ventricular transseptal approach (procedure success rate)
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Procedure
Number analyzed (Participants) | 20
Participants | 20

3. Secondary Outcome: NYHA Class
Description: Improvement in New York Heart Association (NYHA) functional class by >=1 NYHA functional class is a very widely used measure of symptoms in heart failure.
  Improvement is considered to be a decrease in class, representing improve symptoms
  Class Patient Symptoms I No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea (shortness of breath).
  II Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
  III Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  IV Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
Time Frame: Baseline, 6 months
Population: Those patients who attended follow-up at six months were analysed
Measure: Number; unit: participants
Arm/Group | Procedure
Number analyzed (Participants) | 18
participants | 9

4. Secondary Outcome: Number of Participants With >1 Point Improvement in EQ-5D-5L Quality of Life Score
Description: Change in quality of life as measured using the EQ-5D-5L (EuroQol five dimension, five level score ) tool (>1 point decrease)
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number from 1 to 5 that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  Increase in score for each dimension represent worsening of symptoms/ problems
Time Frame: Baseline, 6 months
Population: Those patients who attended follow-up at six months and completed the questionnaires were analysed
Measure: Count of Participants; unit: Participants
Arm/Group | Procedure
Number analyzed (Participants) | 16
Participants | 9

5. Secondary Outcome: Number of Participants With ≥10% Increase in 6-minute Walk Distance
Description: Change in 6 minute walk distance; ≥10% increase
Time Frame: Baseline, 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Procedure
Number analyzed (Participants) | 16
Participants | 10

6. Secondary Outcome: Echocardiographic Response: Change in Ejection Fraction as Measured by Echocardiography From Baseline to 6 Months
Description: Change in echocardiographic parameters of cardiac function ejection fraction was measured using two-dimensional echocardiography and the Simpson method at baseline and six months
Time Frame: Baseline, 6 months
Population: Those patients who attended follow-up at six months and had an echocardiogram with interpretable data were analysed
Measure: Mean (Standard Deviation); unit: % cardiac ejection fraction
Arm/Group | Procedure
Number analyzed (Participants) | 16
% cardiac ejection fraction | 41 (9)

7. Secondary Outcome: Biochemical Response: Change in BNP (B-type Natriuretic Peptide) Levels Between Baseline and Six Months
Description: Change in BNP (b-type natriuretic peptide) levels
  BNP levels were measured from a standard blood draw at baseline and six months.
Time Frame: Baseline, 6 months
Population: Those patients who attended follow-up at six months and had both baseline and six month BNP results available were analysed
Measure: Mean (Standard Deviation); unit: pmol/L
Groups:
- Procedure: 20 patients were recruited, 15 with failed transvenous LV lead placement and 5 non-responders to CRT.
  Baseline BNP (pmol/L) 81 ± 96
Arm/Group | Procedure
Number analyzed (Participants) | 13
pmol/L | 95 (129)

8. Secondary Outcome: Clinical Outcomes
Description: Systemic thrombosis at 2 years
Time Frame: 2 years
Population: Those patients who had follow-up available for any time period more than three months were included
Measure: Count of Participants; unit: Participants
Arm/Group | Procedure
Number analyzed (Participants) | 18
Participants | 3

ADVERSE EVENTS:
Arm/Group | Procedure
All-Cause Mortality (participants affected / at risk) | 3/20
Serious Adverse Events (participants affected / at risk) | 3/18
Other Adverse Events (participants affected / at risk) | 2/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Procedure (N=18)
Stroke or transient ischaemic attack (Nervous system disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Procedure (N=20)
wound haematoma, requiring early re-operation (Injury, poisoning and procedural complications) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes